CLINICAL TRIAL: NCT00080340
Title: Phase 3 Randomized Study of TLK286 (Telcyta) Versus Gefitinib (Iressa) as Third-Line Therapy in Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of TLK286 (Telcyta) vs. Gefitinib in Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Telik (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.3020
Record Dates: First submitted 2004-03-26; First posted 2004-03-30 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2006-03

CONDITIONS: Non Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TER 286; Injections; Gefitinib

INTERVENTIONS:
Drug: TLK286 (Telcyta) HCl for Injection
Drug: gefitinib (Iressa)

SUMMARY:
The purpose of this study is to determine if TLK286(Telcyta) is more effective than gefitinib (Iressa) in the treatment of non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-small cell lung cancer
* Non-small cell lung cancer that is not curable with surgery, radiation, or combined modality chemoradiation
* Failed two prior chemotherapy regimens which must have included platinum
* Measurable disease

Exclusion Criteria:

* Treatment with more than two prior chemotherapy regimens
* History of bone marrow transplantation or stem cell support
* Pregnant or lactating women
* Known history of prior gefitinib therapy
* Known history of prior TLK286 therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520
Dates: Study Completion 2005-05

CONTACTS AND LOCATIONS:
Locations (310):
- United States (242):
  - UAB CCC Clinical Studies Unit, Birmingham, Alabama
  - Department of Veterans Affairs Medical Center, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Little Rock Hematology Oncology Benton, Benton, Arkansas
  - Highlands Oncology Group, Bentonville, Arkansas
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Heritage Physician Group, Oncology, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - East Bay Medical Oncology/Hematology Medical Associates, Inc., Antioch, California
  - East Valley Hematology Oncology Medical Group, Burbank, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - Marilyn Norton, M. D., Chula Vista, California
  - Rosalba Rodriquez, M. D., Chula Vista, California
  - Bay Area Cancer Research Group, Concord, California
  - Wilshire Oncology Medical Group, Inc., Glendora, California
  - Grossmont Hospital, La Mesa, California
  - Sharp Rees-Stealy, La Mesa, California
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - North Valley Hematology Oncology Group, Mission Hills, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - Beverly Oncology & Imaging, Montebello, California
  - Beverly Oncology and Imaging Center, Inc., Montebello, California
  - Clinical Trials & Research Associates, Inc., Montebello, California
  - Oncology Care Medical Associates, Inc., Montebello, California
  - N. County Oncology Medical, Oceanside, California
  - Wilshire Oncology Medical Group, Inc., Pasadena, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - Wilshire Oncology Medical Group, Inc., Rancho Cucamonga, California
  - Southern California Permanente Medical Group, San Diego, California
  - Medical Oncology Associates - SD, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Oncology Care Medical Associates, Inc., San Gabriel, California
  - East Bay Medical Oncology/Hematology Medcial Associates, Inc., San Leandro, California
  - Santa Monica Hematology/Oncology, Santa Monica, California
  - Diablo Valley Oncology & Hematology Medical Group, Inc., Walnut Creek, California
  - Wilshire Oncology Medical Group, Inc., West Covina, California
  - Oncology Care Medical Associates, Inc., Whittier, California
  - Medical Oncology & Hematology, P. C., Hamden, Connecticut
  - Medical Oncology & Hematology, P.C., Meriden, Connecticut
  - Medical Oncology & Hematology, P. C., New Haven, Connecticut
  - New Milford Hospital, New Milford, Connecticut
  - Northwestern Connecticut Oncology/Hematology, New Milford, Connecticut
  - Northwestern Connecticut Oncology/Hematology, Sharon, Connecticut
  - Sharon Hospital, Sharon, Connecticut
  - Charlotte Hungerford Hospital, Torrington, Connecticut
  - Northwestern Connecticut Oncology/Hematology, Torrington, Connecticut
  - Medical Oncology & Hematology, P.C., Waterbury, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Hospital Center - Washington Cancer Institute, Washington D.C., District of Columbia
  - Moroose, Reynolds, Castillo, Robinson & Lukeman, MD, PA, Altamonte Springs, Florida
  - The Center for Hematology/Oncology, Boca Raton, Florida
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Hitesh Patel, Clearwater, Florida
  - Joseph DeFelice, Clearwater, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Oncology Physicians, Clearwater, Florida
  - Space Coast Medical Associates, Cocoa Beach, Florida
  - The Center for Hematology/Oncology, Delray Beach, Florida
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Speicalists, Fort Myers, Florida
  - South Florida Oncology Hematology, Hollywood, Florida
  - Florida Oncology Associates, Jacksonville, Florida
  - Shands Jacksonville, Jacksonville, Florida
  - University of Florida/Jacksonville Faculty Clinic, Jacksonville, Florida
  - Florida Oncology Associates, Jacksonville Beach, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Space Coast Medical Associates, Merritt Island, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Mohammad Kamal, M. D., Ocala, Florida
  - Ocala Research Institute, Inc., Ocala, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Florida Hospital, Orlando, Florida
  - Hematology & Oncology Consultants, PA, Orlando, Florida
  - Moroose, Reynolds, Castillo, Robinson & Lukman, MD, PA, Orlando, Florida
  - Florida Hospital Memorial Division, Cancer Care Center, Ormond Beach, Florida
  - Florida Oncology Associates, Palatka, Florida
  - Palm Beach Cancer Institute, Palm Beach Gardens, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Hematology/Oncology Associates of The Treasure Coast, Port Saint Lucie, Florida
  - Florida Oncology Associates, Saint Augustine, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Palm Beach Cancer Institute, Wellington, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Hematology & Oncology Consultants, PA, Winter Park, Florida
  - Peachtree Hematology & Oncology Consultants, P. C., Atlanta, Georgia
  - Peachtree Hematology & Oncology Consultants, P. C., Fayetteville, Georgia
  - Straub Clinic & Hospital, Honolulu, Hawaii
  - Kapiolani Medical Center for Women & Children, Honolulu, Hawaii
  - North Shore Oncology Hematology Associates, Barrington, Illinois
  - Swedish Covenant Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Central IL, Decatur, Illinois
  - Decatur Memorial Hospital/Clinical Research, Decatur, Illinois
  - Cancer Care Specialists of Central IL, Effingham, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Flossmoor, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - St. Mary Medical Center, Galesburg, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Deerpath Medical Associates, Lake Forest, Illinois
  - North Shore Oncology Hematology Associates, Libertyville, Illinois
  - North Shore Oncology Hematology Associates, McHenry, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Morris, Illinois
  - Hematology Oncology Associates of Illinois (HOAI), Skokie, Illinois
  - Midwest Cancer Research Group, Inc., Skokie, Illinois
  - North Shore Cancer Research Association, Skokie, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer CAre at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Indiana University-Clarian Health Partners, Indianapolis, Indiana
  - Veterans Administration, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana
  - Cancer Care Center, Jeffersonville, Indiana
  - LaPorte Hospital, La Porte, Indiana
  - Medical Consultants, PC, Muncie, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Ball Cancer Center at Forest Ridge Medical Pavilion, New Castle, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph's Regional Medical Center, South Bend, Indiana
  - Medical Center of Vincennes, Vincennes, Indiana
  - Tricare, Vincennes, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Genesis Health System, Davenport, Iowa
  - Kansas City Cancer Center, Kansas City, Kansas
  - Kansas City Cancer Center, Overland Park, Kansas
  - Annapolis Oncology Center, Annapolis, Maryland
  - Auerbach Hematology Oncology Associates, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Associates in Oncology/Hematology, P.C., Kensington, Maryland
  - Associates in Oncology/Hematology, P.C., Rockville, Maryland
  - Department of Hematology/Oncology, Worcester, Massachusetts
  - Fallon Clinic Pharmacy-Linda Tolf, R.Ph., Worcester, Massachusetts
  - Saint Vincent Hospital/Worcester Medical Center-Paul Seed, R.Ph.D, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Cancer Center, OC 139, Ann Arbor, Michigan
  - Sparrow Health System, Lansing, Michigan
  - Lakeland Hospital, Niles, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Duluth Clinic, Duluth, Minnesota
  - Boone Hospital Center, Columbia, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Ellis Fischel Cancer Center - University of Missouri Health Care, Columbia, Missouri
  - Freeman Cancer Institute, Joplin, Missouri
  - Freeman Health System, Joplin, Missouri
  - Kansas City Cancer Center, Kansas City, Missouri
  - Kansas City Cancer Center, Lee's Summit, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Horizons West Medical Group, Scottsbluff, Nebraska
  - Nevada Cancer Centers, Las Vegas, Nevada
  - Central Jersey Oncology Center, East Brunswick, New Jersey
  - University Hospital, Newark, New Jersey
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - New Mexico Oncology Hematology Consultants, Ltd., Albuquerque, New Mexico
  - New York Oncology Hematology, P. C., Albany, New York
  - Business Park Drive, Armonk, New York
  - North Shore Hematology Oncology Associates, P.C., East Setauket, New York
  - Queens Medical Associates, Fresh Meadows, New York
  - New York Oncology Hematology, P.C., Latham, New York
  - Alice Hyde Medical Center, Malone, New York
  - Myrna Sanchez, MD, Malone, New York
  - Albert Einstein Cancer Center at the Montefiore Medical Park, The Bronx, New York
  - The Jack D. Weiler Hospital of the Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Raleigh Hematology Oncology Associates, Cary, North Carolina
  - Raleigh Hematology Oncology Association, Cary, North Carolina
  - Carolinas HealthCare System/Carolinas Medical Center, Charlotte, North Carolina
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Regional Hematology Oncology Associates, Durham, North Carolina
  - Regional Hematology Oncology Association, Durham, North Carolina
  - Gaston Hematology & Oncology Associates, Gastonia, North Carolina
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Raleigh Hematology Oncology Association, Raleigh, North Carolina
  - Piedmont Hematology Oncology Associates, Winston-Salem, North Carolina
  - Cancer Treatment & Research Center, Bismarck, North Dakota
  - Odyssey Research, Bismarck, North Dakota
  - Dakota Cancer Institute, Fargo, North Dakota
  - Odyssey Research, Fargo, North Dakota
  - Case Western Reserve University- University Hospitals of Cleveland, Cleveland, Ohio
  - Mid Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Mid Ohio Oncology/Hematology, Columbus, Ohio
  - Community Health Partners, Ireland Cancer Center, Elyria, Ohio
  - UHHS Chagrin Highlands - Ireland Cancer Center, Orange, Ohio
  - Mid Ohio Oncology/Hematology, Inc., Westerville, Ohio
  - UHHS Westlake - Ireland Cancer Center, Westlake, Ohio
  - Cancer Care Associates, Norman, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Vita Hematology Oncology, P.C., Bethlehem, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Greater Philadelphia Cancer and Hematology Specialists, PC, Philadelphia, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - Medical University of S.C., Charleston, South Carolina
  - Cancer Centers of the Carolinas, Easley, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Cancer Centers of the Carolinas, Greenwood, South Carolina
  - Cancer Centers of the Carolinas, Seneca, South Carolina
  - Cancer Centers of the Carolinas, Spartanburg, South Carolina
  - Chattanooga Oncology & Hemtology Associates, P. C., Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - The Consultant Group, P.C., Franklin, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Gallatin, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Thompson Oncology Group, Knoxville, Tennessee
  - Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - East Tennessee Oncology/Hematology, P.C., Knoxville, Tennessee
  - Baptist Hospital West, Knoxville, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Thompson Oncology Group, Maryville, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - The Consultant Group, P.C., Nashville, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Nashville, Tennessee
  - Cumberland Oncology & Hematology, Oak Ridge, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Dallas Oncology Consultants, PA, Dallas, Texas
  - Center for Oncology Research and Treatment, PA, Dallas, Texas
  - Texas Cancer Associates, LLP, Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Southwest Fort Worth Cancer Center, Fort Worth, Texas
  - The University of Texas - M. D. Anderson Cancer Center, Houston, Texas
  - Center for Oncology Research and Treatment, PA, Richardson, Texas
  - Shore Cancer Center, Nassawadox, Virginia
  - Northwest Medical Specialists, PLLC, Federal Way, Washington
  - Northwest Medical Specialties, PLLC, Lakewood, Washington
  - Northwest Medical Specialists, PLLC, Tacoma, Washington
  - VLCC-Elkhorn, Elkhorn, Wisconsin
  - Medical Consultants, Ltd., Milwaukee, Wisconsin
  - Aurora Health Center-Slinger, Slinger, Wisconsin
  - VLCC-West Bend, West Bend, Wisconsin
- Argentina (13):
  - Policlinica Privada Instituto de Medicina Nuclear, Bahía Blanca, Buenos Aires
  - Instituto Alexander flaming, Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires, Capital Federal, Buenos Aires
  - Hospital de Oncologia Maria Curie, Capital Federal, Buenos Aires
  - Hospital Alvarez, Capital Federal, Buenos Aires
  - Hospital Donacion F. Santojanni, Capital Federal, Buenos Aires
  - Hospital Universitario Austral - Servicio de Oncologia, Pilar, Buenos Aires
  - Hospital Privado de Comunidad, Córdoba, Mar Del Plata
  - Complejo Medico de la Policia Federal Argentina "Churruca-Visca" - Servicio de Oncologia, Buenos Aires
  - Hospital General de Agudos "Carlos G. Durand" - Servicio de Oncologia, Buenos Aires
  - Sociedad de Beneficencia Hospital Italiano, Córdoba
  - Instituto CAICI, Rosario
  - H.I.G.A. Eva Peron, San Martín
- Australia (14):
  - Albury Base Hospital, Albury, New South Wales
  - West Albury Barker's Pharmacy, Albury, New South Wales
  - Department of Medical Oncology-Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Department Of Oncology, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Pharmatel Fresenius Kabi Pty Ltd., West Melbourne, Victoria
  - Murray Valley Private Hospital, Wodonga, Victoria
  - Bankstown Lidcombe Hospital - Department of Medical Oncology, Bankstown
  - Royal Hobart Hospital, Hobart
  - Sir Charles Gairdner Hospital, Nedlands
  - Royal North Shore Hospital-Medical Oncology Dept., St Leonards
  - Border Medical Oncology - Murray Valley Private Hospital, Wodonga
  - Clinical Trials Centre - Wollongong Hospital, Wollongong
- Brazil (17):
  - Instituto do Cancer do Ceara, Fortaleza, Ceará
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Associacao de Combate ao cancer de Goias - Hospital, Goiânia, Goiás
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Hospital das Clinicas da UFPR, Curitiba, Paraná
  - Pro Onco Centro de Tratamento Oncologico S/C Ltda., Curitiba, Paraná
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas-PUCRS, Porto Alegre, Rio Grande do Sul
  - Santo Andre Diagnostico e Tratamento Ltda, Santo André, São Paulo
  - Santo Andre Diagnosticos e Tratamentos Ltda., Santo André, São Paulo
  - Santo Andre Diagnosticos e Tratamentos, Santo André, São Paulo
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo, São Paulo
  - Complexo Hospitalar Heliopolis, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP/EPM, São Paulo, São Paulo
  - Hospital das Clinicas - Universidade de Sao Paulo, São Paulo, São Paulo
  - Fundacao Pio XII - Hospital do Cancer de Barretos, São Paulo, São Paulo
  - Conjunto Hospitalar de Sorocaba, São Paulo, São Paulo
- Chile (9):
  - Departmento de Hemato-Oncologia, Santiago, Las Condes
  - Clinica Las Condes, Santiago
  - Clinica Santa Maria, Santiago
  - FundacionArturo Lopez Perez, Santiago
  - Hospital Clinico Universidad de Chile, Santiago
  - Hospital FACH, Santiago
  - Hospital Militar, Santiago
  - Instituto Nacional del Cancer - Servicio de Radioterapia, Santiago
  - Instituto Nacional del Cancer, Santiago
- Germany (9):
  - Askllepios Fachkliniken, Robert-Koch-Allee 2, Gauting
  - KH GroBhansdorf - Abt. fuer Thoraxonkologie, Woehrendamm 80, Grosshansdorf
  - Laborgemeinschaft Hamburg, Lademannbogen 8, Hamburg
  - Allgemeines Krankenhaus St. Georg, Lohmuehlstr.5, Hamburg
  - St. Vincentius-Kliniken gAG, Sudendstrasse 32, Karlshure
  - Thoraxklinik-Heidelberg GmbH, Heidelberg, Rohrbach BW
  - Stadtisches Krankenhaus Martha-Maria Halle-Dolau GmbH, Haale
  - Allgemeines Kraken Haus St. Georg Onkologie, Hamburg
  - IORC GmbH, Hamburg
- Italy (3):
  - Ospedale Garibaldi di Nesima - Oncologia Medica, Via Palermo, Catania
  - Ospedale "Carlo Poma" - Divisione di Oncologia Medica ed, Via Albertoni, Mantova
  - Azienda Ospedaliera di Parma - U.O. di Oncologia, Parma
- United Kingdom (3):
  - Department of Medical Oncology, West Smithfield, London
  - Bristol Haemotolgy and Oncology Centre, Bristol
  - Div. of cancer Medicine - Princess Alexandra Centre-Ninewells Hospital & Medical School, Dundee

REFERENCES:
- See also: Related Info — http://www.telik.com